CLINICAL TRIAL: NCT03790891
Title: Adoptive Immunotherapy for Non-Hodgkin Lymphoma With CD19-TriCAR-T/SILK Cell
Brief Title: Treatment of Non-Hodgkin Lymphoma With CD19-TriCAR-T/SILK Cell Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Timmune Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-127
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: CAR-T; TriCAR-T; CD19-TriCAR-T; CD19-TriCAR-SILK; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-TriCAR-T/SILK (Experimental): CD19-TriCAR-T/SILK cells will be administered intravenously
  Interventions: Biological: CD19-TriCAR-T/SILK

INTERVENTIONS:
Biological: CD19-TriCAR-T/SILK — A conditioning chemotherapy regimen of fludarabine and cyclophosphamide may be administered, followed by a single infusion of CD19-TriCAR-T cells or 4 repeat infusions of CD19-TriCAR-SILK cells.

SUMMARY:
This is a single arm, open-label, early phase Ⅰ study, to determine the safety and efficacy of CD19-TriCAR-T and CD19-TriCAR-SILK cell therapy in Non-Hodgkin lymphoma treatment.

DETAILED DESCRIPTION:
CD19-TriCAR contains an anti-CD19 scFv, a PD-L1 blocker, and a cytokine complex, enabling the CD19-TriCAR-T/SILK to simultaneously targeting the CD19 positive Non-Hodgkin lymphoma，blocking the inhibitory PD-L1 signal and stimulating innate T/NK cell activation and expansion, thus make it a tri-functional CAR (Tri-CAR). CD19-TriCAR-T is an autologous tri-functional CAR-T cell therapy, CD19-TriCAR-SILK is an Allogeneic tri-functional CAR-NK cell therapy, patients ineligible for leukapheresis or CAR-T therapy will be recommended for CD19-TriCAR-SILK therapy.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must personally sign and date the consent form before initiating any study specific procedures or activities;
2. All subjects must be able to comply with all the scheduled procedures in the study;
3. Refractory or relapsed malignant Non-Hodgkin lymphoma, defined as one or more of the following: Relapsed in 6 months after most recent therapy; Progressive disease in standard chemotherapy; Disease progression or relapsed in ≤12 months of ASCT;
4. At least one measurable lesion per revised IWG Response Criteria;
5. Aged <70 years;
6. Expected survival ≥12 weeks; Eastern cooperative oncology group (ECOG) performance status of≤2;
7. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks;
8. All other treatment induced adverse events must have been resolved to ≤grade 1;
9. Laboratory tests must fulfill the following criteria: ANC ≥ 1000/uL, HGB>70g/L, Platelet count ≥ 50,000/uL, Creatinine clearance ≤1.5 ULN, Serum ALT/AST ≤2.5 ULN, Total bilirubin ≤1.5 ULN (except in subjects with Gilbert's syndrome);

Exclusion Criteria:

1. Presence of fungal, bacterial, viral, or other infection that is hardly to control（defined by investigator）;
2. Patients with symptomatic central nervous system metastasis, intracranial metastasis, and cancer cells found in cerebrospinal fluid are not recommended to participate in this study. Symptom free or post-treatment stable disease or disappearance of lesions should not be excluded. The specific selection is ultimately determined by the investigator;
3. Lactating women or women of childbearing age who plan to conceive during the time period;
4. Active infection with hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive);
5. Known history of infection with HIV;
6. Subjects need systematic usage of corticosteroid;
7. Subjects need systematic usage of immunosuppressive drug;
8. Planed operation, history of other related disease, or any other related laboratory tests restrict patients for the study;
9. Other reasons the investigator consider the patient may not be suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
safety （Incidence of treatment-related adverse events as assessed by CTCAE v4.03） | 24 months
  Incidence of treatment-related adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Complete response rate[CR] (Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma) | 24 months
  Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma
Partial response rate [PR] （Partial response rate per the revised International Working Group (IWG) Response Criteria） | 24 months
  Partial response rate per the revised International Working Group (IWG) Response Criteria
Duration of Response （The time from response to relapse or progression） | 24 months
  The time from response to relapse or progression
Progression Free Survival （The time from the first day of treatment to the date on which disease progresses） | 24 months
  The time from the first day of treatment to the date on which disease progresses
Overall Survival （The number of patient alive, with or without signs of cancer） | 24 months
  The number of patient alive, with or without signs of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yao Hongxia, Principal Investigator — Hainan General Hospital
Locations (3):
- China (3):
  - Hainan Cancer Hospital, Haikou, Hainan
  - Hainan General Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Locke FL, Neelapu SS, Bartlett NL, Siddiqi T, Chavez JC, Hosing CM, Ghobadi A, Budde LE, Bot A, Rossi JM, Jiang Y, Xue AX, Elias M, Aycock J, Wiezorek J, Go WY. Phase 1 Results of ZUMA-1: A Multicenter Study of KTE-C19 Anti-CD19 CAR T Cell Therapy in Refractory Aggressive Lymphoma. Mol Ther. 2017 Jan 4;25(1):285-295. doi: 10.1016/j.ymthe.2016.10.020. Epub 2017 Jan 4. PMID 28129122
- [Background] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994
- [Background] Porter D, Frey N, Wood PA, Weng Y, Grupp SA. Grading of cytokine release syndrome associated with the CAR T cell therapy tisagenlecleucel. J Hematol Oncol. 2018 Mar 2;11(1):35. doi: 10.1186/s13045-018-0571-y. PMID 29499750